CLINICAL TRIAL: NCT00773214
Title: Identification and Characterization of Individual Variability in Exercise-induced Weight Loss: Biological and Behavioral Markers of Success.
Brief Title: Inter Individual Variation in Weight Loss Response to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18926
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Obesity; Appetite; Body composition; Energy compensation
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 12-week supervised exercise programme (5 times /week at 75% maximal Heart Rate)

SUMMARY:
The identification and characterization of individuals who vary in their response to exercise-induced weight loss is important. Weight loss in response to exercise is variable and it remains unknown who will succeed, why, and more importantly how to improve weight loss efficacy.

This study will examine changes in behavioural, metabolic, physiological and biochemical variables in response to a 12 week supervised exercise programme and evaluate their association with weight loss in overweight and obese sedentary individuals.

Our hypothesis is that changes in the plasma levels of appetite related hormones undermine the inter individual variation in weight loss in response to exercise.

This study will improve the understanding of variability to exercise-induced weight loss and allow more individually tailored and appropriate strategies for weight management programmes.

DETAILED DESCRIPTION:
Purpose - To identify predictors of weight loss in overweigh/obese volunteers following a 12 week supervised exercise programme, and to characterise the variability in weight loss response.

Method - Longitudinal study aiming to identify predictors of weight loss in response to a 12-week exercise programme in healthy overweight/obese volunteers.

Subjective and objective measures of appetite, cardiovascular fitness, anthropometry, body composition, resting metabolic rate (RMR), fat and carbohydrate oxidation in the fasting state will be measured at baseline, before participants enroll for the study and after the exercise intervention.

The preload/test-meal paradigm (using a high and low-energy preload: HEP vs LEP) will be used to assess short-term appetite control before and after the exercise intervention following a randomized single-blinded crossover design. Moreover, the long-term effects of exercise on cytokine plasma levels and fasting and postprandial levels of appetite related hormones/metabolites will also be assessed at baseline and end of the study. Participants will act as their own controls throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 25<BMI<35 Kg/m2
* weight stable on the last three months (<2kg)
* not currently dieting to lose weight
* with an inactive lifestyle (not engaged in strenuous work or in regular brisk leisure time exercise more than once a week or in light exercise for more than 20 minutes/day in more than 3 times/week)

Exclusion Criteria:

* History of endocrine/cardiovascular/pulmonary/kidney disease, anaemia, gout, depression or other psychological disorders
* Eating disorders
* Drug or alcohol abuse within the last two years
* Current medication known to affect appetite or induce weight loss.
* Those with a planned surgery during the study period or participating in another research study will also not be accepted to take part in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in fasting and postprandial plasma levels of appetite related hormones | Baseline and after a 12 week exercise intervention

SECONDARY OUTCOMES:
Changes in body weight and body composition | Baseline and after a 12-week exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Catia Martins, BSc, MSc, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Martins C, Kulseng B, King NA, Holst JJ, Blundell JE. The effects of exercise-induced weight loss on appetite-related peptides and motivation to eat. J Clin Endocrinol Metab. 2010 Apr;95(4):1609-16. doi: 10.1210/jc.2009-2082. Epub 2010 Feb 11. PMID 20150577